CLINICAL TRIAL: NCT06775808
Title: Total Infectome Characterization of Eye Infections: a Metagenomic Sequencing Based Observational Study
Brief Title: Total Infectome Characterization of Eye Infections
Status: Recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Fourth People's Hospital Tongji University (Other); The Central Hospital of Huanggang (Other)
Responsible Party: Principal Investigator, Biao Yan, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: SHGH-CRU-2024516
Record Dates: First submitted 2025-01-06; First posted 2025-01-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Eye Infections; Diagnosis
Keywords: infectome; metagenomic sequencing
MeSH Terms: conditions — Eye Infections; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Conjunctival sac swabs (1 swab for each involving eye), intraocular fluid (more than 100μl).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Eye infections cohort: Patients diagnosed with on one or more type of eye infections (including acute conjunctivitis, keratitis, uveitis, and endophthalmitis).

SUMMARY:
Multiple pathogens can cause eye infection. In recent years, emerging and resurging viral infections represent an important public health problem. Many emerging viruses cause infectious diseases involving ophthalmic manifestations, including Mpox virus, Zika, Ebola, and SARS-CoV-2. Broad and unbiased pathogen surveillance is essential, so we design this unbiased metagenomic sequencing based study to investigate the total infectome of eye infections. The study is historical and prospective in design.

DETAILED DESCRIPTION:
This is an investigator-initiated observational study to describe the total infectome of eye infections using metagenomic sequencing. The eye infections, including acute conjunctivitis, keratitis, uveitis, and endophthalmitis, are diagnosed by experienced ophthalmologists according to routine clinical exams.

For the collection of additional biological samples apart from the diagnosis and treatment process, written informed consent is required from the eligible subjects or their legal guardians at the recruitment time is required. The application for exemption of informed consent has been made for using clinical surplus samples. After completing informed consent, subjects will be sampled, and their clinical information will be collected.

Biospecimens, including conjunctival sac swabs (1 swab for each involving eye), or intraocular fluid (more than 100μl), will be collected for metagenomic sequencing using the Illumina NovaSeq X Plus platform.

The clinical information of participants will be collated from electronic medical record information system, including (1) demographic characteristics: age, sex, comorbidities; (2) laboratory examination: blood routine test, immune inflammatory factors, clinical microbiology examination (PCR, serological examination, culture, etc.); (3) imaging examination: anterior segment photograph, corneal endothelial cell examination, corneal confocal microscopy, fundus photograph.

Meta-transcriptomic analysis of the ocular samples will be conducted to identify viruses, bacteria, fungi and parasites. The abundance of pathogens is indicated as the RPKM (i.e. Reads Per Million divided by the length of the reference genome, measured in kilobases).

Eligible participants will be recruited consecutively between August, 2024 and December, 2026 in Department of Ophthalmology, Shanghai General Hospital. The total study duration is expected to be two years from the first subject enrolled to the final analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a clinical diagnosis of one or more types of eye infections (including acute conjunctivitis, keratitis, uveitis, and endophthalmitis).
2. Biological samples has been collected for clinical microbiological examination, or consented to participate in this study.

Exclusion Criteria:

1. Patients who have no historically clinical surplus specimens.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with one or more types of eye infections (including acute conjunctivitis, keratitis, uveitis, and endophthalmitis).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The pathogen profile | through study completion, an average of 2 year
  The bacteria, fungi, viruses, and parasites identified through metagenomic techniques in ocular samples.

SECONDARY OUTCOMES:
Microbial abundance | through study completion, an average of 2 year
  The pathogen abundance is measure by the RPKM (i.e. Reads Per Million divided by the length of the reference genome, measured in kilobases).

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Su, PhD, Study Director — Fudan University
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
IPD could be available on request to the principle investigators.

REFERENCES:
- [Background] Vasquez-Perez A, Magan T, Volpe G, Osborne SF, McFaul K, Vahdani K. Necrotizing Blepharoconjunctivitis and Keratitis in Human Monkeypox. JAMA Ophthalmol. 2023 Mar 1;141(3):285-288. doi: 10.1001/jamaophthalmol.2022.6253. PMID 36757718
- [Background] Rose-Nussbaumer J, Doan T. Role of Ophthalmology in Emerging Infectious Diseases. JAMA Ophthalmol. 2022 Oct 1;140(10):935. doi: 10.1001/jamaophthalmol.2022.4017. PMID 36069833
- [Background] Barshak MB, Durand ML, Gupta A, Mohareb AM, Dohlman TH, Papaliodis GN. State-of-the-Art Review: Ocular Infections. Clin Infect Dis. 2024 Nov 22;79(5):e48-e64. doi: 10.1093/cid/ciae433. PMID 39571607
- [Background] Durand ML, Barshak MB, Sobrin L. Eye Infections. N Engl J Med. 2023 Dec 21;389(25):2363-2375. doi: 10.1056/NEJMra2216081. No abstract available. PMID 38118024
- [Background] Ranjan R, Ranjan S. Ocular Pathology: Role of Emerging Viruses in the Asia-Pacific Region-A Review. Asia Pac J Ophthalmol (Phila). 2014 Sep-Oct;3(5):299-307. doi: 10.1097/APO.0000000000000021. PMID 26107917
- [Background] Tsui E, Sella R, Tham V, Kong AW, McClean E, Goren L, Bahar I, Cherian N, Ramirez J, Hughes RE Jr, Privratsky JK, Onclinx T, Feit-Leichman R, Cheng A, Molina I, Kim P, Yu C, Ruder K, Tan A, Chen C, Liu Y, Abraham T, Hinterwirth A, Zhong L, Porco TC, Lietman TM, Seitzman GD, Doan T; SCORPIO Study Group. Pathogen Surveillance for Acute Infectious Conjunctivitis. JAMA Ophthalmol. 2023 Dec 1;141(12):1140-1144. doi: 10.1001/jamaophthalmol.2023.4785. PMID 37917077
- [Background] Austin A, Lietman T, Rose-Nussbaumer J. Update on the Management of Infectious Keratitis. Ophthalmology. 2017 Nov;124(11):1678-1689. doi: 10.1016/j.ophtha.2017.05.012. Epub 2017 Sep 21. PMID 28942073
- [Background] Ai JW, Weng SS, Cheng Q, Cui P, Li YJ, Wu HL, Zhu YM, Xu B, Zhang WH. Human Endophthalmitis Caused By Pseudorabies Virus Infection, China, 2017. Emerg Infect Dis. 2018 Jun;24(6):1087-1090. doi: 10.3201/eid2406.171612. PMID 29774834
- [Background] Wu F, Zhao S, Yu B, Chen YM, Wang W, Song ZG, Hu Y, Tao ZW, Tian JH, Pei YY, Yuan ML, Zhang YL, Dai FH, Liu Y, Wang QM, Zheng JJ, Xu L, Holmes EC, Zhang YZ. A new coronavirus associated with human respiratory disease in China. Nature. 2020 Mar;579(7798):265-269. doi: 10.1038/s41586-020-2008-3. Epub 2020 Feb 3. PMID 32015508
- [Background] Chiu CY, Miller SA. Clinical metagenomics. Nat Rev Genet. 2019 Jun;20(6):341-355. doi: 10.1038/s41576-019-0113-7. PMID 30918369
- [Background] Burton MJ, Ramke J, Marques AP, Bourne RRA, Congdon N, Jones I, Ah Tong BAM, Arunga S, Bachani D, Bascaran C, Bastawrous A, Blanchet K, Braithwaite T, Buchan JC, Cairns J, Cama A, Chagunda M, Chuluunkhuu C, Cooper A, Crofts-Lawrence J, Dean WH, Denniston AK, Ehrlich JR, Emerson PM, Evans JR, Frick KD, Friedman DS, Furtado JM, Gichangi MM, Gichuhi S, Gilbert SS, Gurung R, Habtamu E, Holland P, Jonas JB, Keane PA, Keay L, Khanna RC, Khaw PT, Kuper H, Kyari F, Lansingh VC, Mactaggart I, Mafwiri MM, Mathenge W, McCormick I, Morjaria P, Mowatt L, Muirhead D, Murthy GVS, Mwangi N, Patel DB, Peto T, Qureshi BM, Salomao SR, Sarah V, Shilio BR, Solomon AW, Swenor BK, Taylor HR, Wang N, Webson A, West SK, Wong TY, Wormald R, Yasmin S, Yusufu M, Silva JC, Resnikoff S, Ravilla T, Gilbert CE, Foster A, Faal HB. The Lancet Global Health Commission on Global Eye Health: vision beyond 2020. Lancet Glob Health. 2021 Apr;9(4):e489-e551. doi: 10.1016/S2214-109X(20)30488-5. Epub 2021 Feb 16. No abstract available. PMID 33607016